CLINICAL TRIAL: NCT05005338
Title: An Open Label Phase 1 Study to Determine the Absolute Bioavailability of Single and Repeated Daily Oral Administration of BIIB122 (DNL151) Utilizing a Microtracer Dose of Intravenously Administered [14C] BIIB122 ([14C] DNL151) to Healthy Subjects
Brief Title: A Study to Determine the Absolute Bioavailability of BIIB122/DNL151 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 283HV103
Record Dates: First submitted 2021-07-27; First posted 2021-08-13 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — DNL151

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort A (Experimental)
  Interventions: Drug: BIIB122 (DNL151); Drug: [14C] BIIB122 ([14C] DNL151)

INTERVENTIONS:
Drug: BIIB122 (DNL151) — Oral doses
Drug: [14C] BIIB122 ([14C] DNL151) — Intravenous doses

SUMMARY:
This is a single center, non-randomized, open label Phase 1 study to determine the PK and absolute bioavailability of BIIB122 (DNL151) in 2 conditions: following a single, oral dose of BIIB122 (DNL151) and following consecutive days of oral dosing, approximating steady state.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Women of non-childbearing potential and men either with a vasectomy, using contraception, or having sex with a woman of non-childbearing potential
* Body mass index (BMI) ≥ 18 kg/m2 and ≤ 32 kg/m2
* Considered to be in good health
* Nonsmoker

Key Exclusion Criteria:

* History or presence of any condition or prior surgery that, in the opinion of the investigator, poses a significant risk to subject safety and/or achievement of study objectives

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
PK Parameter: The first time to maximum observed concentration (Tmax) of BIIB122 (DNL151) in plasma following oral administration | 1 day
PK Parameter: Maximum observed concentration (Cmax) of BIIB122 (DNL151) in plasma following oral administration | 1 day
PK Parameter: Area under the concentration-time curve (AUC) of BIIB122 (DNL151) and [14C]-BIIB122 ([14C]-DNL151 in plasma following oral and intravenous administration | 1 day
PK Parameter: Time from baseline at which half of BIIB122 (DNL151) and [14C]-BIIB122 ([14C]-DNL151 has been eliminated (t1/2) in plasma after oral and intravenous administration | 1 day
PK Parameter: Clearance (CL/F and CL) of BIIB122 (DNL151) and [14C]-BIIB122 ([14C]-DNL151) from plasma after oral and intravenous administration | 1 day
PK Parameter: Volume of distribution (Vd/F and Vd) of BIIB122 (DNL151) and [14C]-BIIB122 ([14C]-DNL151) from plasma after oral and intravenous administration | 1 day
PK Parameter: Absolute bioavailability (F) of BIIB122 (DNL151) after oral administration | 1 day
PK Parameter: The first time to maximum observed concentration (Tmax) of BIIB122 (DNL151) in plasma following oral administration | 21 days
PK Parameter: Maximum observed concentration (Cmax) of BIIB122 (DNL151) in plasma following oral administration | 21 days
PK Parameter: Concentration of BIIB122 (DNL151) in plasma at the end of dosing interval | 21 days
PK Parameter: Area under the concentration-time curve of BIIB122 (DNL151) and [14C]-BIIB122 ([14C]-DNL151) in plasma following oral and intravenous administration | 21 days
PK Parameter: Time from baseline at which half of BIIB122 (DNL151) and [14C]-BIIB122 ([14C]-DNL151) has been eliminated (t1/2) in plasma after oral and intravenous administration | 21 days
PK Parameter: Volume of distribution (Vd/F and Vd) of BIIB122 (DNL151) and [14C]-BIIB122 ([14C]-DNL151) from plasma after oral and intravenous administration | 21 days
PK Parameter: Clearance (CL/F and CL) of BIIB122 (DNL151) and [14C]-BIIB122 ([14C]-DNL151) from plasma after oral and intravenous administration | 21 days
PK Parameter: Absolute bioavailability (F) of BIIB122 (DNL151) after oral administration | 21 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 31 days
Incidence of serious adverse events (SAEs) | 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Denali Therapeutics Inc.
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No